CLINICAL TRIAL: NCT05514418
Title: Viral Non-Suppression, Drug Resistance, Perceptions and Effectiveness of Intensive Adherence Counselling Among People Living With HIV/AIDS on Antiretroviral Therapy With Low-Level Viraemia in Uganda.
Brief Title: Effectiveness of Intensive Adherence Counselling Among People Living With HIV/AIDS With Low-level Viraemia in Uganda.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Makerere University (Other)
Collaborators: Rakai Health Sciences Project (Unknown); Ministry of Health, Uganda (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SPH-2021-144
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This group will receive three monthly sessions of intensive adherence counselling (IAC) and psychosocial support, using the 5 A's principles for chronic care (which include; Assess, Advise, Agree, Assist and Arrange). Each monthly IAC session will be offered by the research assistants for about one hour, and adherence will also be assessed by pill counts. Colour-coded IAC forms will be developed and used to differentiate the study from routine IAC services for the non-suppressed patients; and the study will be conducted on different days, from those on which the routine clinic occurs.
  Following the three months of the study, all the study participants both in the control and intervention groups will be reviewed at the health facility and a repeat viral load (VL) test done for each of the participants, to determine whether they have achieved a non-detectable VL or not.
  Interventions: Procedure: Intensive Adherence Counselling (IAC)
- Control Arm (No Intervention): This group will comprise of participants who will receive the routine standard of care. These participants will receive the normal patient education and encouragement to continue with their antiretroviral therapy (ART) at the start of the study. They will not be reviewed monthly or offered any counselling for the entire three months. These participants will be given an appointment after three months for repeat viral load (VL) testing.

INTERVENTIONS:
Procedure: Intensive Adherence Counselling (IAC) — Intensive adherence counselling is offered to people living with HIV (PLHIV) having a non-suppressed viral load (VL) result ( a VL of 1,000 copies/ml or more) and this is given once every month for three months. In our study, we are going to give IAC to PLHIV with low-level viraemia (having a VL of 50 copies/ml but less than 1,000 copies/ml) and determine its effectiveness in causing a non-detectable VL (less than 50 copies/ml), which is desirable for PLHIV on ART.
  Other Names: Targeted Adherence Counselling; Enhanced Adherence Counselling
  Arms: Intervention Arm

SUMMARY:
Uganda uses a threshold of 1,000 copies/ml to determine HIV viral non-suppression among people living with HIV/AIDS (PLHIV) on treatment, which is indicative of either poor adherence or HIV virologic treatment failure; as per the recent WHO recommendations. The use of this high threshold of 1,000 copies/ml has resulted into an increase in the number of PLHIV having low-level viraemia (≥50 to <1,000 copies/ml) from 11.0% in 2017 to 35.0% in 2020 in Uganda. Different studies in developed countries have shown that low-level viraemia is associated with HIV drug resistance, and despite this, there is no intervention to manage and control low-level viraemia (LLV), as per the recent Uganda national HIV guidelines. With this increasing and unmanaged low-level viraemia (LLV), Uganda might never achieve the global targets of ending AIDS as epidemic by 2030, as stipulated by target 3.3 of SDG 3.

This study will therefore determine the effectiveness of intensive adherence counselling on achieving a non-detectable viral load (below 50 copies/ml) in the management of LLV among PLHIV on ART in Uganda. This study will generate useful information that might guide the review of the national HIV guidelines, to control and manage LLV among PLHIV on ART; and thereby enable Uganda to achieve the global goals of SDG 3, Target 3.3 and the national targets of Vision 2040.

DETAILED DESCRIPTION:
Study design This study will be a cluster randomized clinical trial, which will determine the effectiveness of IAC in achieving a non-detectable viral load among PLHIV on ART with LLV from selected health facilities from all the four regions of Uganda. The outcome of the study will be the proportions of PLHIV with a non-detectable viral load in both the intervention and control arms of the study.

Study setting The study will be conducted in selected health facilities from each of the four regions in Uganda (Central, Eastern, Northern and Western).

Study population The study will comprise of PLHIV on ART who have had recent VL result with LLV.

Sample size A sample size of 79 participants per arm will be estimated from; n = [(Zα/2 + Zβ)2 × {(p1 (1-p1) + (p2 (1-p2))}]/(p1 - p2)2 (Sakpal, 2010; Sullivan, 2020); with a power of 90% and a 5% level of significance to detect a 15% difference in PLHIV on ART who get a non-detectable viral load between those offered IAC and those who are not. IAC is an intervention used to manage PLHIV with a non-suppressed VL and 70% of these PLHIV attain viral suppression (WHO, 2016); and therefore, we assume that p2 is 0.7. PLHIV with LLV have suppressed VL and we assume IAC to even be more effective at about 90% in creating a non-detectable VL in these PLHIV, hence we assume p1 to be 0.9.

An equal sample size of 12 participants for each of the 8 clusters will be estimated from (Hemming et al., 2011) where nI is the number of participants required for each arm, k is the number of clusters, and p is the intra-cluster correlation estimate, which is 0.0180 (Barnhart et al., 2016), thus a total of 96 participants is required. Considering a design effect of 1.126 and an attrition rate of 20%, the resultant total sample size of 136 participants per study arm will be used, hence a total 17 participants will be recruited per cluster.

Sampling procedure The clusters will be grouped into pairs based on the geographical location (Lorenz et al., 2018). In each cluster pair, one cluster will be randomly assigned to the intervention arm, which will receive intensive adherence counselling (IAC) as an intervention to manage LLV. Hence both the intervention and control arms will be balanced.

Data collection The study will take place at the HIV clinics of the selected health facilities (clusters), and the selected research assistants who will either be ART counsellors or clinicians or nurses will be oriented and trained about the study and also re-mentored in how to offer IAC sessions.

PLHIV on ART with recent VL results having LLV who will have consented to take part in the study will sequentially be recruited into the clusters, and the demographic data will be collected.

Control Arm (Standard of Care): This arm will comprise of clusters which will receive the routine standard of care. These participants in these clusters will receive the normal patient education and encouragement to continue with their ART at the start of the study. They will not be reviewed monthly or offered any counselling for the entire three months. These participants will be given an appointment after three months for repeat VL testing.

Intervention Arm (IAC arm): The participants of clusters in this arm will receive three monthly sessions of intensive adherence counselling and psychosocial support, using the 5 A's principles for chronic care (which include; Assess, Advise, Agree, Assist and Arrange). Each monthly IAC session will be offered by the research assistants for about one hour, and adherence will also be assessed by pill counts. Colour-coded IAC forms will be developed and used to differentiate the study from routine IAC services for the non-suppressed patients; and the study will be conducted on different days, from those on which the routine clinic occurs.

Following the three months of the study, all the study participants in all the clusters both in the control and intervention arms will be reviewed at the health facility and a repeat VL done for each of the participants, to determine whether they have achieved a non-detectable VL or not.

Statistical Analysis EpiData version 3.02 will be used for data entry, and analysis will be done using Stata version 14. Descriptive statistics will be used to describe the sample size. The proportions of PLHIV attaining a non-detectable VL in the intervention arm will be compared with those PLHIV attaining a non-detectable VL in the control arm. The effectiveness of intensive adherence counselling will be estimated using Cox regression models, adjusted for sociodemographic factors.

ELIGIBILITY:
Inclusion Criteria:

* People living with HIV (PLHIV) on antiretroviral therapy (ART) with recent viral load (VL) results having low-level viraemia (≥50 to <1,000 copies/ml)
* PLHIV aged 18 years or above

Exclusion Criteria:

* Critically sick PLHIV
* Non-suppressed PLHIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-02-12 (Estimated); Study Completion 2023-04-12 (Estimated)

PRIMARY OUTCOMES:
Proportions of people living with HIV (PLHIV) with a non-detectable viral load (below 50 copies/ml) in both the intervention and control arms of the study | 3 completed months of IAC
  Number of people living with HIV (PLHIV) with a non-detectable viral load (below 50 copies/ml) in both the intervention and control arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Nicholus Nanyeenya, MBChB, MPH, Principal Investigator — Makerere University
Locations (8):
- Uganda (8):
  - Kamuli General Hospital, Jinja
  - Kiyunga health centre IV, Jinja
  - Mityana General Hospital, Kampala
  - Mpigi Health Centre IV, Kampala
  - Alebtong health centre IV, Lira
  - Orum health centre IV, Lira
  - Rwekubo health centre IV, Mbarara
  - TASO Mbarara, Mbarara

IPD SHARING:
Plan to Share IPD: No
No plan to share the IPD yet

REFERENCES:
- [Derived] Nanyeenya N, Nakanjako D, Makumbi F, Nakigozi G, Nalugoda F, Kigozi G, Nasuuna E, Kibira SPS, Nabadda S, Kiyaga C, Huzaifah M, Kiwanuka N. Effectiveness of intensive adherence counselling in achieving an undetectable viral load among people on antiretroviral therapy with low-level viraemia in Uganda. HIV Med. 2024 Feb;25(2):245-253. doi: 10.1111/hiv.13568. Epub 2023 Oct 18. PMID 37853605